CLINICAL TRIAL: NCT00183430
Title: Prazosin for Noncombat Trauma PTSD
Brief Title: Prazosin for Treating Noncombat Trauma Post-Traumatic Stress Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH069867 (NIH); R01MH069867 (NIH); DATR AD-TS
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Post-Traumatic Stress Disorder; Sleep Initiation and Maintenance Disorders
Keywords: Prazosin; Sleep Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Prazosin; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive treatment with prazosin plus psychotherapy
  Interventions: Drug: Prazosin; Behavioral: Psychotherapy
- 2 (Placebo Comparator): Participants will receive treatment with placebo plus psychotherapy
  Interventions: Drug: Placebo; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Prazosin — Prazosin capsules 1 to 25 mg are taken orally twice per day in divided doses at 10 am and bedtime.
  Other Names: Minipress
  Arms: 1
Drug: Placebo — Placebo capsules are taken orally twice per day at 10 am and bedtime.
  Arms: 2
Behavioral: Psychotherapy — All participants will undergo psychotherapy during medication treatment period.

SUMMARY:
This study will evaluate the effectiveness of prazosin in treating post-traumatic stress disorder caused by noncombat trauma in individuals taking selective serotonin reuptake inhibitors.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is an anxiety disorder that can develop after exposure to a terrifying event in which grave physical harm occurred or was threatened. People with PTSD have persistent frightening thoughts and memories of their past ordeal and often feel emotionally numb, especially with people to whom they were once close. PTSD was first recognized in male combat veterans. Today, however, the majority of people who have PTSD are young women who have experienced non combat-related trauma, such as sexual or physical assault or a life-threatening illness or accident. The disorder can be short-lived, but PTSD can also become chronic, with long lasting symptoms that are often treatment-resistant, possibly causing severe functional disability. Frequent trauma-related nightmares and other debilitating sleep disruptions are examples of chronic PTSD symptoms for which an effective treatment has not been developed. Sertraline and paroxetine, both selective serotonin reuptake inhibitors (SSRIs), are the only drugs approved by the FDA for treating PTSD. Neither of them, however, has been effective in reducing PTSD-related sleep disruption. Studies have shown that the drug prazosin has been effective in reducing distressing trauma-related nightmares in older male combat veterans. This study will evaluate the effectiveness of prazosin in treating post-traumatic stress disorder caused by noncombat trauma in individuals already being treated with SSRIs.

Participants in this double-blind study will first undergo 12 weeks of treatment with psychotherapy and a standard SSRI. After 12 weeks, participants will be randomly assigned to receive either prazosin or placebo in addition to psychotherapy and standard SSRI treatment for a total of 8 weeks. Study visits will occur weekly for the first 12 weeks, and then at Weeks 1, 2, 4, 6, and 8 during the 8-week phase. Additionally, follow-up visits will be held 4 and 18 weeks post-intervention. PTSD symptoms, disorder severity, and frequency of sleep disturbances will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of PTSD, as derived from the Clinician-Administered PTSD Scale (CAPS)
* Stabilized on any necessary medications for at least 4 weeks prior to study entry
* Score of greater than 4 on the CAPS Recurrent Distressing Dreams item (maximum score of 8)
* Score of greater than 4 on the CAPS Difficulty Falling or Staying Asleep item (maximum score of 8)
* Agrees to use an effective form of contraception throughout the study

Exclusion Criteria:

* Any acute or significant chronic medical illness
* Any unstable medical condition
* Unstable angina, recent heart attack, history of congestive heart failure, pre-existing hypotension (systolic blood pressure less than 110 mm Hg), or orthostatic hypotension
* Insulin-dependent diabetes
* Chronic kidney or liver failure
* Pancreatitis or gout
* Meniere's disease, benign positional vertigo, or narcolepsy
* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist
* Currently taking another alpha-1 antagonist agent
* Pregnant
* DSM-IV diagnosis of cognitive disorder, schizophrenia, schizoaffective disorder, bipolar disorder, or other psychotic disorder
* Current delirium
* Active substance dependence disorder within 3 months of study entry
* Current substance use other than alcohol (no more than 2 drinks per day)
* Severe psychiatric instability or situational life crises, including evidence of suicidal or homicidal ideation
* Currently taking any other psychotropic medication (e.g., antidepressants, benzodiazepines, anti-convulsants, anti-psychotics, sedating antihistamines, sedatives/hypnotics (exclusionary medications will be discontinued and participants will undergo a 2-week washout period before baseline assessments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-10; Primary Completion 2009-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray A. Raskind, MD, Principal Investigator — University of Washington/Department of Veterans Affairs
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Raskind MA, Peskind ER, Kanter ED, Petrie EC, Radant A, Thompson CE, Dobie DJ, Hoff D, Rein RJ, Straits-Troster K, Thomas RG, McFall MM. Reduction of nightmares and other PTSD symptoms in combat veterans by prazosin: a placebo-controlled study. Am J Psychiatry. 2003 Feb;160(2):371-3. doi: 10.1176/appi.ajp.160.2.371. PMID 12562588
- [Background] Raskind MA, Thompson C, Petrie EC, Dobie DJ, Rein RJ, Hoff DJ, McFall ME, Peskind ER. Prazosin reduces nightmares in combat veterans with posttraumatic stress disorder. J Clin Psychiatry. 2002 Jul;63(7):565-8. doi: 10.4088/jcp.v63n0705. PMID 12143911
- [Background] Raskind MA, Dobie DJ, Kanter ED, Petrie EC, Thompson CE, Peskind ER. The alpha1-adrenergic antagonist prazosin ameliorates combat trauma nightmares in veterans with posttraumatic stress disorder: a report of 4 cases. J Clin Psychiatry. 2000 Feb;61(2):129-33. doi: 10.4088/jcp.v61n0208. PMID 10732660
- [Background] Peskind ER, Bonner LT, Hoff DJ, Raskind MA. Prazosin reduces trauma-related nightmares in older men with chronic posttraumatic stress disorder. J Geriatr Psychiatry Neurol. 2003 Sep;16(3):165-71. doi: 10.1177/0891988703256050. PMID 12967060
- [Background] Taylor FB, Martin P, Thompson C, Williams J, Mellman TA, Gross C, Peskind ER, Raskind MA. Prazosin effects on objective sleep measures and clinical symptoms in civilian trauma posttraumatic stress disorder: a placebo-controlled study. Biol Psychiatry. 2008 Mar 15;63(6):629-32. doi: 10.1016/j.biopsych.2007.07.001. Epub 2007 Sep 14. PMID 17868655
- [Background] Raskind MA, Peskind ER, Hoff DJ, Hart KL, Holmes HA, Warren D, Shofer J, O'Connell J, Taylor F, Gross C, Rohde K, McFall ME. A parallel group placebo controlled study of prazosin for trauma nightmares and sleep disturbance in combat veterans with post-traumatic stress disorder. Biol Psychiatry. 2007 Apr 15;61(8):928-34. doi: 10.1016/j.biopsych.2006.06.032. Epub 2006 Oct 25. PMID 17069768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from April 2002 through July 2008. Participants were recruited from VA outpatient clinics and flyers in the community.
Pre-assignment Details: no significant events.
Groups:
- Prazosin: Participants will receive treatment with prazosin plus psychotherapy
  Prazosin : Prazosin capsules 1 to 25 mg are taken orally twice per day in divided doses at 10 am and bedtime.
  Psychotherapy : All participants will undergo psychotherapy during medication treatment period.
- Placebo: Participants will receive treatment with placebo plus psychotherapy
  Placebo : Placebo capsules are taken orally twice per day at 10 am and bedtime.
  Psychotherapy : All participants will undergo psychotherapy during medication treatment period.
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 9 | 11
Completed | 3 | 11
Not Completed | 6 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — did not meet inclusion criteria | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11.6) | 46 (9.4) | 44 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression of Change
Description: The Clinical Global Impression of Change is a 7-point scale that rates global change compared to baseline (1=markedly improved, 2=moderately improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=moderately worse, 7=markedly worse). The Clinical Global Impression of Change is used to determine the impact of treatment effects on meaningful and distinct change in overall sense of well-being and functioning. This outcome measure evaluates change from Baseline to Week 8.
Time Frame: Baseline to Week 8
Population: Number of participants analyzed equals the number of participants who were able to complete this assessment at Week 8.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 3 | 11
Units on a Scale | 2.33 (0.58) | 3.27 (0.90)

2. Primary Outcome: Change in Recurring Distressing Dreams and Difficulty Falling and Staying Asleep Items of the CAPS
Description: Item B-2 "recurrent distressing dreams of the event" is a single item from teh Clinician Administered PTSD Scale (CAPS). The rating consists of two parts: Frequency plus Intensity. Symptom frequency rated 0 to 4. Symptom intensity rated 0 to 4. Frequency plus Intensity ratings equal the total score. The total minimum score = zero. The total maximum score = 8. A higher score is worse; a lower score is better. This outcome measure evaluates the change in score from Baseline to Week 8.
Time Frame: Baseline to Week 8
Population: Number of participants analyzed equals the number of participants who were able to complete this assessment at Week 4.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 3 | 11
Units on a Scale | -2.00 (.82) | -1.09 (1.93)

3. Primary Outcome: Change in Sleep Assessed by the Pittsburgh Sleep Quality Index
Description: Pittsburgh Sleep Quality Index is a self-report questionnaire assessing sleep quality and disturbances over a 1-month time interval. A global score is obtained by summing the seven component subscales (total score range: 0-21). A score of 5 or less indicates good sleep quality. A score of more than 5 indicates poor sleep quality. Change is measured from Baseline to Week 8.
Time Frame: Baseline to Week 8
Population: Number of participants analyzed equals the number of participants who were able to complete this assessment at Week 8.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 3 | 11
Units on a Scale | 4 (0.82) | 2.09 (4.42)

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning at Baseline (initiation of study drug) through Week 8.
Arm/Group | Prazosin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/11
Other Adverse Events (participants affected / at risk) | 2/3 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Prazosin (N=3) | Placebo (N=11)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
migraine headache (Vascular disorders) | 1 (2) | 0 (0)
presyncope episodes (General disorders) | 1 (2) | 0 (0)
sinusitis (General disorders) | 1 (1) | 0 (0)
adverse drug reaction (not study drug) (General disorders) | 1 (2) | 0 (0)
Spider Bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
strep throat (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1/1 (1) | 4 (5)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
elevated energy and mood (Psychiatric disorders) | 0 (0) | 1 (1)
chest pain consistent with dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
conjunctivitis (Eye disorders) | 0 (0) | 1 (2)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Decreased ability to urinate (Renal and urinary disorders) | 0 (0) | 1 (1)
dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
fibroclastic breast disease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
herpes simplex 1 outbreak (Infections and infestations) | 0 (0) | 1 (1)
increased sadness (Psychiatric disorders) | 0 (0) | 1 (1)
metacarpophalangeal inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
edema (General disorders) | 0 (0) | 1 (1)
menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 1 (1)
panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
paroxysmal nocturnal dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
protinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
calf muscle soreness (General disorders) | 0 (0) | 1 (1)
sciatic nerve pain (Nervous system disorders) | 0 (0) | 1 (1)
sinus congestion (General disorders) | 0 (0) | 1 (1)
sinus infection (Infections and infestations) | 0 (0) | 1 (1)
ulnar nerve transposition (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No